CLINICAL TRIAL: NCT05025774
Title: Fitness and Lung Function Among Survivors of Heart Transplant, Leukemia and Infant Bronchopulmonary Dysplasia (BPD, Also Known as Chronic Lung Disease of Prematurity) Through Exercise (FLASHLITE)
Brief Title: Fitness and Lung Function Among Survivors of Heart Transplant, Leukemia and Infant BPD Through Exercise
Acronym: FLASHLITE
Status: Recruiting | Type: Observational
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: PEDS-2021-29482
Record Dates: First submitted 2021-08-05; First posted 2021-08-27 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Chronic Lung Disease; Chronic Obstructive Pulmonary Disease; Acute Lymphoblastic Leukemia; Heart Transplant
Keywords: Quality of life; Lung function; Fitness; Exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample specimens will be saved for future use investigating biomarkers and/or Blood will be drawn from each participant and then separated and frozen as serum and mononuclear cells. Samples will be stored in the Department of Pediatrics freezers on the University of Minnesota Twin Cities campuses. All samples will be labeled with a unique participant ID number and no personal or identifiable data. Samples will be maintained for up to 5 years. Planned analysis include biomarker assessments. Samples will only be accessible to individuals listed on the IRB approval for this study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Adolescent or young adult acute lymphoblastic leukemia survivor, OR living with chronic lung disease of prematurity, OR living with heart transplant
  Interventions: Other: Physical activity
- Control: 14-25 years old healthy individuals who are ambulatory without assistance. We may enroll younger subjects but we wish to subjects to match our patient population
  Interventions: Other: Physical activity

INTERVENTIONS:
Other: Physical activity — Participant Reported Physical Activity and Outcomes (completed via REDCap or on paper)

SUMMARY:
This study aims to more accurately assess cardiac function, ventilation and exercise capacity in a non-invasive fashion, and to better characterize exercise intolerance in the setting of three populations of individuals with chronic diseases of childhood (acute lymphoblastic leukemia (ALL), chronic lung disease (CLD) of prematurity, and post-heart transplant (HT))

DETAILED DESCRIPTION:
Physical activity in childhood is an integral part of maintaining health and quality of life. Children who participate in routine physical activity are more likely to maintain a healthy body weight and are less likely to have heart disease, type 2 diabetes and high blood pressure as adults. Children with chronic disease are often limited from full participation in exercise for various reasons -perceived physical limitations, either from the patient and family or from their medical provider, or because of symptoms which cause exercise to feel uncomfortable. As the number of children living and aging with chronic disease continues to grow, the researchers are hoping to expand the current exercise testing capabilities for both clinical care and research in order to (i) provide data to permit formulation of evidence-based guidelines for exercise in chronic childhood disease; (ii) improve understanding of limitations to exercise in this growing population; (iii) learn long-term implications of chronic childhood disease as these individuals enter adulthood.

ELIGIBILITY:
Inclusion Criteria:

* Cases:

  * Acute lymphoblastic leukemia survivor, OR living with chronic lung disease of prematurity, OR living with heart transplant
  * 8-25 years old
  * Height: ≥ 48 inches
  * Ambulatory without assistance
  * English speaking
  * Normotensive (<95th percentile for age; okay if managed with antihypertensive medication)
  * SpO2 >92%
  * Not pregnant
  * ALL survivor specific: must have completed therapy ≥ 3 months prior to study entry
* Controls

  * 8-25 years old
  * Height: ≥ 48 inches
  * Ambulatory without assistance
  * English speaking
  * No history of arrhythmia or known cardiac dysfunction at baseline
  * Normotensive (<95th percentile for age; okay if managed with antihypertensive medication)
  * SpO2 >95%
  * Not pregnant

Exclusion Criteria:

* Cases:

  * ALL specific: received cranial radiation, bone marrow transplant recipients
  * Investigator or patient's primary physician deems the patient unsuitable for the study
* Controls:

  * History of malignancy, CLD or HT or any other diagnosis which may reduce cardiorespiratory function
  * Investigator deems the patient unsuitable for the study

Ages: 8 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: The case participants are the ALL survivors, CLD due to prematurity patients, and post-HT recipients. The control participants can be medical students, UMN staff's children, UMN/Fairview staff, medical residents and undergraduate or graduate students. The remaining controls will be from other UMMCH clinics with conditions unlikely to impact exercise capacity such as dermatology, orthopedics or sports medicine and the University Children's Clinic. Approval will be granted from the treating physician before approaching the control participants
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Measure of Peak O2 intake during test exercise | 3-4 hours during the onetime study visit day
  Maximal cardiopulmonary exercise testing (CPX) will be completed on cycle ergometer to determine peak oxygen uptake, a measure of cardiorespiratory fitness
Measure of Cardiac output during test exercise | 3-4 hours during the onetime study visit day
  Cardiac output is measured using C2H2 open-circuit breathing technique: a mass spectrometer medical gas analyzer will measure gas concentration continuously, yielding serial Stroke Volume measurements during incremental exercise. Cardiac output is the product of heart rate and stroke volume

SECONDARY OUTCOMES:
The proportion of expiratory flow limitation (EFL) | 3-4 hours during the onetime study visit day
  The proportion of expiratory flow limitation (EFL) during exercise while tracking dyspnea and perceived exertion
Association between cardiac function and patient reported outcomes of perceived fitness | 3-4 hours during the onetime study visit day
  Logistic regression will be used to understand associations between cardiac function and patient reported outcomes of perceived fitness

CONTACTS AND LOCATIONS:
Overall Officials: Pianosi Paolo, MD, Principal Investigator — Masonic Children's Hospital, University of Minnesota
Locations (1):
- Masonic Cancer Center, Minneapolis, Minnesota, United States